CLINICAL TRIAL: NCT03701828
Title: Liver Health and Metabolic Function in People With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201808128
Record Dates: First submitted 2018-09-10; First posted 2018-10-10 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Bariatric Surgery; Anastomosis, Roux-en-Y; Biliopancreatic Diversion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Weight loss (Experimental): Participants will undergo weight loss surgery
  Interventions: Procedure: Weight loss surgery

INTERVENTIONS:
Procedure: Weight loss surgery — All surgery types will be included. However, only participants scheduled for surgery with collaborating surgeons will be included. Surgery is not provided by study team.
  Other Names: Sleeve gastrectomy, Roux-en-Y, biliopancreatic diversion

SUMMARY:
This project aims to determine the effect of significant weight loss on rates on hepatic fibrogenesis in people with obesity.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) affects approximately 70% of those with obesity and if left untreated can progress to cirrhosis and liver failure. NAFLD stages progress from the stage of simple steatosis to steatohepatitis, and fibrosis The stage of NAFLD is currently best determined using histology from a liver biopsy, however this provides a static depiction of the state of the liver. Therefore, this project aims to determine fibrogenesis in the liver of obese humans in vivo, before and after weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥35 kg/m2
* Scheduled for Bariatric surgery

Exclusion Criteria:

* Significant organ disfunction/disease
* Tobacco use
* Previous bariatric surgery
* Pregnancy
* Excessive alcohol use
* Liver disease other than NAFLD

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-02-19 (Actual)

PRIMARY OUTCOMES:
Liver histology | Before and after ~20% weightloss, up to 6 months
  Analysis of liver tissue morphology
Hepatic Fibrogenesis | Before and after ~20% weightloss, up to 6 months
  Rates of liver collagen synthesis

SECONDARY OUTCOMES:
Plasma protein synthesis | Before and after ~20% weightloss, up to 6 months
  Synthesis rates of collagen-related proteins in plasma
Tissue inflammation | Before and after ~20% weightloss, up to 6 months
  adipose tissue and blood immune cell content
Systemic inflammation | Before and after ~20% weightloss, up to 6 months
  Plasma cytokine concentrations
Body composition | Before and after ~20% weightloss, up to 6 months
  Body composition assessed by dual-energy x-ray absorptiometry and magnetic resonance scans
Adipose histology | Before and after ~20% weightloss, up to 6 months
  Assessment of adipose tissue morphology
Tissue gene expression | Before and after ~20% weightloss, up to 6 months
  Messenger ribonucleic acid content of adipose, liver and blood tissues will be assessed
Tissue lipidomics | Before and after ~20% weightloss, up to 6 months
  bioactive lipid content of adipose, liver and blood tissues will be assessed
Insulin sensitivity | Before and after ~20% weightloss, up to 6 months
  Whole-body insulin sensitivity during a hyperinsulinemic-euglycemic clamp
tissue extracellular vesicles | Before and after ~20% weightloss, up to 6 months
  amount, content and function of extracellular vesicles obtained from adipose, liver, and blood tissue
adipose tissue progenitor cells | Before and after ~20% weightloss, up to 6 months
  content and function of progenitor cells obtained from adipose tissue
Liver single cell RNA seq | at the time of surgery only
  gene expression of liver immune cell types
Liver flow cytometry | at the time of surgery only
  liver immune cell content
Liver lipid turnover | Before and after ~20% weightloss, up to 6 months
  Turnover rates of fatty acids and triglycerides
PNPLA3 synthesis | At the time of surgery only
  Synthesis rate of liver PNPLA3 protein

OTHER OUTCOMES:
PNPLA3 genotype | Screening only
  genotyping for the PNPLA3 SNP rs738409 will be determined

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States